CLINICAL TRIAL: NCT06573827
Title: The Urinary Microbiome and Its Relationship to the Urinary and Serum Metabolome in Healthy Peri- and Postmenopausal Women
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: MB-001; 24/RVO-FNOs/2024 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Urinary Tract Infections
Keywords: microbiome; urinary metabolome; urinary bladder; menopause
MeSH Terms: conditions — Urinary Tract Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Microbiome in healthy volunteers: Healthy volunteers willing to provide blood and urine samples for microbiome evaluation
  Interventions: Diagnostic Test: Blood and urine sample evaluation

INTERVENTIONS:
Diagnostic Test: Blood and urine sample evaluation — Blood and urine sample evaluation will be performed in healthy female volunteers.

SUMMARY:
The presented project aims to characterize the microbiome of healthy peri- and postmenopausal women and its correlation with the metabolome of urine and serum.

DETAILED DESCRIPTION:
At the beginning of their visit to the Blood Center of the University Hospital Ostrava, blood and plasma donors will be approached by one of the authorized members of the team with information about the possibility of participating in this study. The course of the study will be explained to them in detail, including the sampling methodology, their processing, and further handling. If the subject is interested in participating in the study, they will give written informed consent to participate in the study. Subsequently, the inclusion and exclusion criteria for participation in the study will be verified. If these are not met, the subject will be excluded from the study. Furthermore, the criteria for current valid blood and urine sampling will be verified. If the conditions for valid sampling are not met and the participant is still interested in participating in the study, she will be offered a new sampling date. If the study subject fulfills the conditions of valid sampling, she will fill out a simple questionnaire, which will be used to obtain data on basic demographic characteristics. Their knowledge is essential for the correct interpretation of urine and serum test results. Blood and serum will then be collected. In justified cases, sampling can also be carried out at the Urology Department of the University Hospital Ostrava. After submitting the first sample, the participant will be asked to submit another urine and serum sample in 3-6 months. By submitting the 2nd urine and serum sample, the participant ends her participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women over 50 years old
* Consent to participate in the study
* Willingness to take urine and blood samples according to the protocol

Exclusion Criteria:

* Known congenital developmental defects of the urinary tract (congenital hydronephrosis, vesicoureteral reflux, renal agenesis, and hypoplasia, multicystic and polycystic kidneys)
* Recurrent urinary tract infections (more than 3 episodes in the last 12 months)
* Presence of any lower-urinary tract symptoms (urgency, frequency, incontinence, stranguria, urge to urinate, weak urine stream, the feeling of post-micturition residue)
* The presence of a foreign body in the urinary tract - urolithiasis, urinary catheter, ureteral stent
* Acute or chronic diseases with possible influence on lower-urinary tract function
* Medications with possible influence on lower-urinary tract function
* Rheumatoid arthritis
* Diabetes mellitus

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only peri- and post-menopausal female probands will be enrolled in the study.
Study Population: Healthy peri- and post-menopausal female volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome alpha-diversity | 6 months
  The number of bacterial species in the urine sample will be assessed.
Microbiome beta-diversity | 6 months
  Inter-individual variability in the proportion of bacterial species will be assessed.

SECONDARY OUTCOMES:
Correlation of microbiome alpha-diversity and serum metabolome | 6 months
  The correlation of microbiome alpha-diversity and serum metabolome will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Krhut, prof.,MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

REFERENCES:
- [Background] Cho I, Blaser MJ. The human microbiome: at the interface of health and disease. Nat Rev Genet. 2012 Mar 13;13(4):260-70. doi: 10.1038/nrg3182. PMID 22411464
- [Background] Turnbaugh PJ, Ley RE, Hamady M, Fraser-Liggett CM, Knight R, Gordon JI. The human microbiome project. Nature. 2007 Oct 18;449(7164):804-10. doi: 10.1038/nature06244. PMID 17943116
- [Background] Monsen T, Ryden P. Flow cytometry analysis using sysmex UF-1000i classifies uropathogens based on bacterial, leukocyte, and erythrocyte counts in urine specimens among patients with urinary tract infections. J Clin Microbiol. 2015 Feb;53(2):539-45. doi: 10.1128/JCM.01974-14. Epub 2014 Dec 3. PMID 25472486
- [Background] Mueller ER, Wolfe AJ, Brubaker L. Female urinary microbiota. Curr Opin Urol. 2017 May;27(3):282-286. doi: 10.1097/MOU.0000000000000396. PMID 28234750
- [Background] Morand A, Cornu F, Dufour JC, Tsimaratos M, Lagier JC, Raoult D. Human Bacterial Repertoire of the Urinary Tract: a Potential Paradigm Shift. J Clin Microbiol. 2019 Feb 27;57(3):e00675-18. doi: 10.1128/JCM.00675-18. Print 2019 Mar. PMID 30404941
- [Background] Salabura A, Luniewski A, Kucharska M, Myszak D, Dolegowska B, Ciechanowski K, Kedzierska-Kapuza K, Wojciuk B. Urinary Tract Virome as an Urgent Target for Metagenomics. Life (Basel). 2021 Nov 19;11(11):1264. doi: 10.3390/life11111264. PMID 34833140
- [Background] Nelson DE, Dong Q, Van der Pol B, Toh E, Fan B, Katz BP, Mi D, Rong R, Weinstock GM, Sodergren E, Fortenberry JD. Bacterial communities of the coronal sulcus and distal urethra of adolescent males. PLoS One. 2012;7(5):e36298. doi: 10.1371/journal.pone.0036298. Epub 2012 May 11. PMID 22606251
- [Background] Antunes-Lopes T, Vale L, Coelho AM, Silva C, Rieken M, Geavlete B, Rashid T, Rahnama'i SM, Cornu JN, Marcelissen T; EAU Young Academic Urologists (YAU) Functional Urology Working Group. The Role of Urinary Microbiota in Lower Urinary Tract Dysfunction: A Systematic Review. Eur Urol Focus. 2020 Mar 15;6(2):361-369. doi: 10.1016/j.euf.2018.09.011. Epub 2018 Sep 28. PMID 30270128
- [Background] Colella M, Topi S, Palmirotta R, D'Agostino D, Charitos IA, Lovero R, Santacroce L. An Overview of the Microbiota of the Human Urinary Tract in Health and Disease: Current Issues and Perspectives. Life (Basel). 2023 Jun 30;13(7):1486. doi: 10.3390/life13071486. PMID 37511861
- [Background] Bar N, Korem T, Weissbrod O, Zeevi D, Rothschild D, Leviatan S, Kosower N, Lotan-Pompan M, Weinberger A, Le Roy CI, Menni C, Visconti A, Falchi M, Spector TD; IMI DIRECT consortium; Adamski J, Franks PW, Pedersen O, Segal E. A reference map of potential determinants for the human serum metabolome. Nature. 2020 Dec;588(7836):135-140. doi: 10.1038/s41586-020-2896-2. Epub 2020 Nov 11. PMID 33177712
- [Background] Lee-Sarwar KA, Lasky-Su J, Kelly RS, Litonjua AA, Weiss ST. Metabolome-Microbiome Crosstalk and Human Disease. Metabolites. 2020 May 1;10(5):181. doi: 10.3390/metabo10050181. PMID 32369899